CLINICAL TRIAL: NCT05017103
Title: A Phase II Clinical Trial Evaluating the Efficacy and Safety of Sintilimab for Advanced Rare Cancers (SiARa Cancer Study) - Undifferentiated Pleomorphic Sarcoma (SiARa-UPS)
Brief Title: Sintilimab for the Treatment of Locally Advanced, Metastatic, Recurrent, or Unresectable Undifferentiated Pleomorphic Sarcoma, SiARa Cancer Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The drug sponsor stopped supporting study.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1046; NCI-2021-08589 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1046 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-10

CONDITIONS: Locally Advanced Undifferentiated Pleomorphic Sarcoma; Metastatic Undifferentiated Pleomorphic Sarcoma; Recurrent Undifferentiated Pleomorphic Sarcoma; Unresectable Undifferentiated Pleomorphic Sarcoma
MeSH Terms: conditions — Histiocytoma, Malignant Fibrous | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (sintilimab) (Experimental): Patients receive sintilimab IV over 30-60 minutes on day 1. Cycles repeat every 3 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Sintilimab

INTERVENTIONS:
Biological: Sintilimab — Given IV
  Other Names: Anti-PD-1 Monoclonal Antibody IBI308; Anti-PDCD1 Monoclonal Antibody IBI308; IBI 308; IBI308

SUMMARY:
This phase II trial investigates the effects of sintilimab in treating patients with undifferentiated pleomorphic sarcoma that has spread to nearby tissue or lymph nodes (locally advanced), spread to other places in the body (metastatic), come back (recurrent), or cannot be removed by surgery (unresectable). Immunotherapy with monoclonal antibodies, such as sintilimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of sintilimab in subjects with undifferentiated pleomorphic sarcoma (UPS) (overall response rate [ORR] at 12 weeks [12W] by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1).

SECONDARY OBJECTIVE:

I. To evaluate the ORR (RECIST 1.1) and disease control rate (DCR), PFS, overall survival (OS), safety and duration of response (DOR) of sintilimab in subjects with UPS.

EXPLORATORY OBJECTIVES:

I. To evaluate the correlation between biomarkers in tumor tissue and efficacy, including but not restricted to PD-L1 expression level, tertiary lymphoid structures (TLS) transcriptome sequencing, single-cell sequencing, and multicolor immunohistochemistry (IHC) analyses.

II. To evaluate the correlation between biomarkers in peripheral blood and efficacy, including but not restricted to soluble PD-L1, circulating tumor deoxyribonucleic acid (DNA) (ctDNA), identification/quantification of immunologic changes, and cytokine analyses.

OUTLINE:

Patients receive sintilimab intravenously (IV) over 30-60 minutes on day 1. Cycles repeat every 3 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 60 days for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed unresectable, locally advanced, recurrent or metastatic UPS
* Refractory or intolerant to at least one line of systemic chemotherapy. Patient ineligible for cytotoxic chemotherapy are eligible
* Aged >= 18
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Subject must be unsuitable for definitive treatment, such as definitive chemoradiotherapy and/or surgery
* Could provide archival or fresh tissues for correlative analysis
* Have at least one measurable lesion as per RECIST version (v)1.1
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L

  * Note: Subjects cannot receive blood transfusion, erythropoietin (EPO), or granulocyte-colony stimulating factor (GSF) within 7 days prior to the blood collection
* Platelet (PLT) count >= 75 x 10^9/L

  * Note: Subjects cannot receive blood transfusion, erythropoietin (EPO), or granulocyte-colony stimulating factor (GSF) within 7 days prior to the blood collection
* Hemoglobin (HGB) >= 8.0 g/dL

  * Note: Subjects cannot receive blood transfusion, erythropoietin (EPO), or granulocyte-colony stimulating factor (GSF) within 7 days prior to the blood collection
* Total bilirubin (TBIL) =< 1.5 x upper limit of normal (ULN) and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x upper limit of normal (ULN) in subjects without hepatic metastasis
* TBIL =< 1.5 x ULN and ALT and AST =< 5 x ULN in subjects with hepatic metastasis. Exception: Patients with known Gilbert disease: serum bilirubin level =< 3 x ULN
* Urine protein < 2+ from random sample or < 1 g from 24-hour urine collection, and creatinine clearance rate (Ccr) >= 60 mL/min by Cockcroft-Gault formula
* Adequate coagulation function, defined as international normalized ratio (INR) =< 1.5 or prothrombin time (PT) =< 1.5 x ULN; if the subject is receiving anticoagulant therapy, the results of coagulation tests need to be within the acceptable range for anticoagulants
* Expected survival >= 12 weeks
* Subject (female subjects of childbearing age or male subjects whose partners are of childbearing age) must take effective contraceptive measures during the entire course of the trial and until 180 days after the last dose
* Signed the informed consent form (ICF) and be able to comply with the scheduled follow-up visits and related procedures required in the protocol

Exclusion Criteria:

* Received treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug that specifically targets T-cell co-stimulation or immune checkpoint pathways
* Enrolled in another interventional clinical study, unless only involved in an observational study (non-interventional) or in the follow-up phase of an interventional study
* Received palliative therapy for local lesion within 2 weeks prior to the first dose
* Received systemic treatment with anti-cancer indications or immunomodulators (including thymosins, interferons, and interleukins) within 2 weeks prior to the first dose of study treatment
* Received systemic immunosuppressants within 2 weeks prior to first dose, excluding local use of glucocorticoids administered by nasal, inhaled, or other routes, and systemic glucocorticoids at physiological doses (no more than 10 mg/day of prednisone or equivalents), or glucocorticoids to prevent allergies to contrast media
* Received a live attenuated vaccine within 4 weeks prior to the first dose of study treatment or be scheduled to receive live attenuated vaccine during the study period.

  * Note: Seasonal inactivated influenza virus vaccines within 4 weeks prior to the first dose of study treatment are permitted, but attenuated influenza vaccines are not
* Received major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of study treatment or is scheduled to receive major surgery during the course of the trial
* Any toxicity (excluding alopecia, events that are not clinically significant, or asymptomatic laboratory abnormalities) due to prior anti-tumor therapy that has not yet resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 grade 0 or 1 prior to the first dose of study treatment
* Known symptomatic central nervous system (CNS) metastasis or carcinomatous meningitis. Subjects with brain metastases who have received prior treatment can be enrolled if the disease is stable (no imaging evidence of progressive disease (PD) for at least 4 weeks prior to the first dose of study treatment), there is no evidence of new brain metastases or progression of the existing metastatic lesion(s) upon repeated imaging, and corticosteroids have not been required for at least 14 days prior to the first dose of study treatment. Patients with carcinomatous meningitis are ineligible, regardless of whether the disease is clinically stable or not
* Subjects with bone metastases at risk of paraplegia
* Known active autoimmune disease requiring treatment or previous disease history within 2 years (subjects with vitiligo, psoriasis, alopecia, or Graves' disease not requiring systemic treatment, hypothyroidism only requiring thyroid replacement, or type I diabetes only requiring insulin can be enrolled)
* Known history of primary immunodeficiency diseases
* Known active pulmonary tuberculosis
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
* Human immunodeficiency virus (HIV)-infected subjects (positive anti-HIV antibody)
* Active or poorly controlled serious infections
* Symptomatic congestive heart failure (New York Heart Association [NYHA] class II-IV) or symptomatic or poorly controlled arrhythmia
* Uncontrolled hypertension (systolic blood pressure >= 160 mmHg or diastolic blood pressure >= 100 mmHg) despite of standard treatment
* Any arterial thromboembolic event within 6 months prior to enrollment, including myocardial infarction, unstable angina, cerebrovascular accident, or transient cerebral ischemic attack
* Significant malnutrition, such as those requiring continuous parenteral nutrition >= 7 days; excluding those having received intravenous treatment for malnutrition for more than 4 weeks before the first dose of study treatment
* History of clinically significant deep venous thrombosis, pulmonary embolism, or other serious thromboembolic events within 3 months prior to enrollment (implantable port or catheter-related thrombosis or incidental PE detected on scan without symptoms or superficial venous thrombosis are not considered as "serious" thromboembolisms)
* Uncontrolled metabolic disorders, non-malignant organ or systemic diseases, or cancer-related secondary diseases that may lead to higher medical risks and/or survival evaluation uncertainties
* Hepatic encephalopathy, hepatorenal syndrome, or cirrhosis with Child-Pugh class B or C
* Bowel obstruction or history of the following diseases: inflammatory bowel disease, extensive bowel resection (partial colectomy or extensive small intestine resection accompanied with chronic diarrhea), Crohn's disease, or ulcerative colitis
* Known acute or chronic active hepatitis B (positive hepatitis B surface antigen [HBsAg] and hepatitis B virus [HBV] DNA viral load >= 104 copies/mL or > 2000 IU/mL), or acute or chronic active hepatitis C (hepatitis C virus [HCV] ribonucleic acid [RNA] > 103 copies/mL), or simultaneously positive for HBsAg and HCV antibody
* History of gastrointestinal (GI) perforation and/or fistula within 6 months prior to the enrollment, excluding gastrostomy or enterostomy
* Interstitial lung disease requiring corticosteroids
* History of other primary malignant tumors, excluding:

  * Malignant tumors that achieved a complete response (CR) at least 2 years prior to enrollment and expected to require no treatment during the trial
  * Adequately treated nonmelanoma skin cancer or lentigo maligna with no sign of disease recurrence
  * Adequately treated carcinoma in situ with no sign of disease recurrence
  * Prostate, chronic lymphocytic leukemia (CLL) or other cancers where the indolent nature of tumor allows for and patient is cancer under active surveillance
* Pregnant or breastfeeding female subjects
* Acute or chronic diseases, psychiatric disorders, or laboratory abnormalities that may lead to the following consequences: increased investigational drug-related risks, interference with interpretation of trial results or considered ineligible for participating in the trial by the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Somaiah, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Sintilimab)
Started | 6
Completed | 4
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Sintilimab)
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate
Description: Will be defined as the proportion of subjects with a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v.1.1) in the evaluable population.
Time Frame: At 12 weeks
Population: 2 participants not evaluable at 12 weeks (passed away)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sintilimab)
Number analyzed (Participants) | 4
Participants
  Progressive Disease | 3
  Stable Disease | 1

ADVERSE EVENTS:
Time Frame: Up to 9 months plus 90 days
Arm/Group | Treatment (Sintilimab)
All-Cause Mortality (participants affected / at risk) | 4/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sintilimab) (N=6)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (6)
Spinal fracture (Musculoskeletal and connective tissue disorders) | 1 (6)
Febrile neutropenia (General disorders) | 1 (6)
Colitis (Gastrointestinal disorders) | 1 (6)
Disease progression (General disorders) | 1 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT05017103/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT05017103/ICF_001.pdf